CLINICAL TRIAL: NCT05479084
Title: Does Kinesio Taping Affect Shooting Performance Acutely in Archery Athletes?
Brief Title: The Effects of Kinesio Taping in Archery
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Eylül Pınar KISA, Lecturer, Biruni University
Other Study IDs: Archery
Record Dates: First submitted 2022-07-26; First posted 2022-07-29 (Actual); Last update posted 2023-01-03 (Actual); Status verified 2022-09

CONDITIONS: Sports Physical Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Kinesiotaping — Kinesio taping will be applied on the lower part of the trapezius.

SUMMARY:
The aim of the study is to investigate the effects of KT on archery athletes' performance.

DETAILED DESCRIPTION:
Archery is a sport that requires strength, endurance, stabilization, and coordination of the upper body and shoulder girdle muscles. Kinesio taping (KT), which increased in popularity with the use in the athletes in the 2008 summer Olympics, is commonly investigated in the literature. KT is claimed to reduce pain and edema, increase functional performance, joint position sense, and blood-lymph flow, provide stability, and improve range of motion, flexibility, and strength. The aim of the study is to investigate the effects of KT on archery athletes' performance.

ELIGIBILITY:
Inclusion Criteria:

* To be archery in the elite category for at least 1 year
* Attending training sessions at least 2 days a week

Exclusion Criteria:

* Having any neurological problems
* Having a Turkish-speaking and reading disability

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Archery athletes
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Assessment of Archery Shooting Performance | 15 minutes
  The archery shooting performance will be assessed with the target paper which includes 5 scoring colors. The subject will be placed within 18 meters distance of the target paper. The subjects will have 12 arrows to make the shoot. The best 6 shoots will be taken to calculate the total score.

SECONDARY OUTCOMES:
Assessment of Proprioception | 15 minutes
  The proprioception will be assessed with the angle reproduction test.
Evaluation of Scapular Dyskinesis | 5 minutes
  Dyskinesis will be assessed with scapular lateral slide test.

CONTACTS AND LOCATIONS:
Overall Officials: Eylül Pınar Kısa, PhD, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No